CLINICAL TRIAL: NCT00004407
Title: Randomized Study of Intravenous Immunoglobulin (IVIg) in Patients With Subacute Proximal Diabetic Neuropathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: 199/13294; MAYOC-91596; MAYOC-FDR001358
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-01

CONDITIONS: Diabetic Neuropathies
Keywords: diabetic amyotrophy; diabetic lumbosacral radiculoplexus neuropathy; diabetic neuropathy; diabetic proximal neuropathy; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Diabetic Neuropathies; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Immunoglobulins

INTERVENTIONS:
Drug: immune globulin

SUMMARY:
OBJECTIVES: I. Determine the effect of intravenous immunoglobulin on recovery time of patients with proximal diabetic neuropathy.

II. Determine whether rate of response is dose dependent in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled study. Patients are randomized to treatment with low dose intravenous immunoglobulin (IVIg), high dose IVIg, or placebo.

Patients must first complete baseline evaluation. Patients receive IVIg or placebo on days 1, 2, 3, and 5, biweekly at weeks 2-4, weekly at weeks 5-8, and every other week at weeks 9-12.

Patients are assessed at 6, 12, 36, 52, and 104 weeks.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnostically proven non-insulin dependent diabetes mellitus as defined by the following criteria: Presence of classic symptoms, such as polyuria, polydipsia, ketonuria, and rapid weight loss, together with plasma glucose elevations Elevated fasting glucose concentration on more than one occasion
* Diagnostically proven proximal diabetic neuropathy with any of the following symptoms: Severe thigh, hip, or leg pain Greater than 20% weight loss Progressive proximal weakness in the painful leg Weakness in the contralateral lower limb Thoracic or cervical root distribution Symmetric distal polyneuropathy or autonomic neuropathy may be mild or absent

--Prior/Concurrent Therapy--

* At least 6 months since prior immunosuppression or plasma exchange
* No history of prior renal transplant

--Patient Characteristics--

* Age: 18 and over
* Performance status: Gait impairment at least grade 2
* Hematopoietic: Not specified
* Hepatic: Not specified
* Renal: Creatinine no greater than 1.4 mg/dL (women) Creatinine no greater than 1.5 mg/dL (men) No history of renal failure
* Cardiovascular: No history of cardiac failure
* Neurologic: Normal nerve conduction studies or changes compatible with distal symmetric diabetic neuropathy or diabetic lumbosacral radioplexus neuropathy Spinal fluid cell count less than 5 cells/mm3 Normal cerebral spinal fluid cytology No structural spine disease No inherited neuropathy
* Other: Electromyographic evidence of proximal lower limb plexus OR Radicular denervation compatible with proximal diabetic neuropathy No other systemic disease or malignancy Normal IgA levels No chronic inflammatory demyelinating polyradiculoneuropathy (CIDP) No systemic amyloidosis No monoclonal gammopathy associated neuropathy No history of allergy to serum products No selective cervical or root involvement without lower limb weakness No evidence of secondary diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 1998-02; Study Completion 2000-03

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J. Windebank, Study Chair — Mayo Clinic